CLINICAL TRIAL: NCT04038554
Title: Microbiota in Acute Pancreatitis: Prospective Multicenter Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Maria Nieves García-Monforte, Senior doctor of Hepatobiliopancreatic Surgery department, Corporacion Parc Tauli
Other Study IDs: CSPT-CG-MPA
Record Dates: First submitted 2019-06-18; First posted 2019-07-31 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Acute Pancreatitis; Microbial Colonization
MeSH Terms: conditions — Pancreatitis; Communicable Diseases | interventions — Defecation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Qualitative and quantitative description of bacterial species present in feces and saliva samples from patients diagnosed with acute pancreatitis of different grades and etiologies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Pancreatitis: Patients older than 18 years old diagnosed of acute pancreatitis according to Atlanta 2012.
  Interventions: Diagnostic Test: Feces and saliva analysis
- Healthy Control: Healthy people with a proximity relationship with case patients and similar age (+/- 5 years).
  Interventions: Diagnostic Test: Feces and saliva analysis

INTERVENTIONS:
Diagnostic Test: Feces and saliva analysis — Qualitative and quantitative analysis of the microbiota in the feces and saliva by mRNA sequencing.

SUMMARY:
The objective of the study is to classify and carry out a quantitative analysis of the different bacterial species present in the intestinal microbiota of patients with acute pancreatitis and determine if there are significant differences regarding healthy controls. At the same time, the investigators pretend to determine if there are differences according to the etiology and severity of the disease and if the disregulation is temporary or is maintained after one month of discharge.

To carry out this purpose, the investigators have designed a prospective and multicentre observational study where samples of feces and saliva of patients admitted for acute pancreatitis of different etiologies and severity will be analyzed.

DETAILED DESCRIPTION:
The study of the human microbiota is gaining importance given its relationship with the homeostasis of the organism as well as with certain pathologies. Specifically in the case of acute and chronic pancreatitis, recent studies suggest the disregulation of the intestinal flora as a possible determinant in the development and evolution of the disease. If this hypothesis is confirmed, hygienic-dietetic measures, as well as the administration of antibiotics, probiotics or fecal transplantation, may have therapeutic implications.

The objective of the study is to classify and carry out a quantitative analysis of the different bacterial species present in the intestinal microbiota of patients with acute pancreatitis and determine if there are significant differences regarding healthy controls. At the same time, the investigators also intend to determine if there are differences according to the etiology and severity of the disease and if the disregulation is temporary or is maintained after one month of discharge.

To carry out this purpose, it has been designed a prospective and multicentre observational study where samples of feces and saliva of patients admitted for acute pancreatitis of different etiologies and severity will be analyzed .

ELIGIBILITY:
Inclusion Criteria:

* Case patients: adult patients diagnosed of acute pancreatitis according to Atlanta 2012 criteria
* Healthy controls: healthy people with a proximity relationship with case patients and similar age (+/- 5 years. Doesn't have to be a parental relationship.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old diagnosed of acute pancreatitis according to Atlanta 2012 criteria with no etnia, gender or comorbilities restriction.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of different microbiological taxonomic groups in fecal and salival samples determined by mRNA sequencing and PCR amplification (Microbiota Composition). | Two determinations: at recruitment and after one month of discharge.
  Assessment of the different number of microbiological taxonomic groups and the proportion of them in fecal and salival samples from patients with acute pancreatitis by mRNA sequencing and PCR amplification using Illumina sequency techonology.

SECONDARY OUTCOMES:
Microbiota composition with respect to pancreatitis etiology assessed by clinical history and complementary tests. | Two determinations: at recruitment and after one month of discharge.
  Assessment of the different number of microbiological taxonomic groups and the proportion of them in fecal and salival samples from patients with different etiology of acute pancreatitis by mRNA sequencing and PCR amplification using Illumina sequency techonology.
  The pancreatitis etiology will be defined according to clinical history (e.g alcohol consumption, cholelitiasis, metabolic and inmune disorders) and complementary tests (US, CT scan and blood tests).
Microbiota composition with respect to pancreatitis severity | Two determinations: at recruitment and after one month of discharge.
  Microbiota composition with respect to pancreatitis severity according to Atlanta 2012 criteria

CONTACTS AND LOCATIONS:
Overall Officials: MNieves García-Monforte, PhD, Principal Investigator — Corporacion Sanitaria Parc Tauli; Robert Memba Ikuga, PhD, Principal Investigator — Fundacion Instituto de Investigacion Pere i Virgili
Locations (2):
- Spain (2):
  - Corporacion Sanitaria Parc Taulí, Sabadell, Barcelona
  - Fundación Instituto de Investigación Pere i Virgili, Tarragona